CLINICAL TRIAL: NCT04939662
Title: Phase II, Single-arm Study of Olaparib and Bevacizumab Combination Therapy in Relapsed Small Cell Lung Cancer Subjects With DNA Damage Response and the Repair Pathway Alteration, ATM Deficiency, SLFN11 Positive, or POU2F3 Positive
Brief Title: Olaparib and Bevacizumab in Relapsed Small Cell Lung Cancer Subjects
Acronym: SUKSES-B2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Se-Hoon Lee (Other)
Collaborators: AstraZeneca (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Se-Hoon Lee, Samsung Medical Center, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUKSES-B2
Record Dates: First submitted 2021-06-02; First posted 2021-06-25 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: SCLC; olaparib; bevacizumab; relapsed small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Interventional Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib+Bevacizumab to SCLC patients (Experimental): Regimen and administration:
  Administration of olaparib Olaparib 300 mg bid per os every 12 hours D1-21 administered in each cycle days. One cycle consists of 21 days. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Administration of bevacizumab Bevacizumab 15 mg/kg via IV administered on Day1 of each cycle. One cycle is consisted of 21 days.
  The subject's body weight criterion is based on C1D1 (first dose date), and if more than 10% of BW is increased and decreased, the drug dose is changed to that BW.
  Interventions: Drug: Olaparib+Bevacizumab to SCLC patients

INTERVENTIONS:
Drug: Olaparib+Bevacizumab to SCLC patients — Olaparib 300 mg bid per os every 12 hours D1-21 administered in each cycle days. One cycle consists of 21 days.
  Bevacizumab 15 mg/kg via IV administered on Day1 of each cycle. One cycle is consisted of 21 days.
  The subject's body weight criterion is based on C1D1 (first dose date), and if more than 10% of BW is increased and decreased, the drug dose is changed to that BW.
  Other Names: Drug Combination Intervention

SUMMARY:
This study is a single arm, multi-centre phase II study of olaparib and bevacizumab combination therapy in subjects with relapsed small cell lung cancer (SCLC) as a second or third line (systemic) therapy.

Subjects will receive olaparib and bevacizumab combination therapy. The arm is composed of 28 subjects.

Olaparib 300 mg bid per os every 12 hours administered each cycle day and bevacizumab 15 mg/kg via IV administered on Day 1 of every cycle for every 3 weeks. One cycle consists of 21 days.

DETAILED DESCRIPTION:
Study design This study is a single arm, multi-centre phase II study of olaparib and bevacizumab combination therapy in subjects with relapsed small cell lung cancer (SCLC) as a second or third line (systemic) therapy.

Subjects will receive olaparib and bevacizumab combination therapy. The arm is composed of 28 subjects.

Olaparib 300 mg bid per os every 12 hours administered each cycle day and bevacizumab 15 mg/kg via IV administered on Day 1 of every cycle for every 3 weeks. One cycle consists of 21 days.

Tumour evaluation by RECIST v1.1 using CT or MRI scans of chest, abdomen, pelvis and brain (optional in case of brain metastases), CEA, NSE and LDH will be conducted at screening (within 28 days prior to first dose of Cycle1 Day1) and every 6 weeks (±1 week) for the first 42 weeks relative to the start of combination therapy (Cycle 1 Day 1), and thereafter every 9 weeks (±1week) until objective disease progression.

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Subjects may continue olaparib and bevacizumab beyond progression (according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a subjects discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Assessments for survival should be made every 3months following objective disease progression. The details of first and subsequent therapies for cancer, after discontinuation of olaparib and bevacizumab treatment, will be collected.

The imaging modalities used for RECIST 1.1 assessment will be CT or MRI scans of chest, abdomen and pelvis. And CEA, NSE and LDH tests are also used for the evaluation. RECIST 1.1 scans will be analysed by the investigator on site.

Subjects may also be requested to provide tumour samples from the primary or metastatic tumours on progression to understand resistance mechanisms. Sample provision is optional and depend on the subject's will.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. SCLC that satisfies one or more of the following conditions; Histologically confirmed SCLC with documented

1) ATM deficiency, SLFN11 positive, POU2F3 positive by immunohistochemistry 2) HR(homologous recombination) pathway gene mutation: BRCA 1/2, MRE11A, BLM, NBN, RAD50, RAD52, RAD54L, RAD51, RAD51B, RAD51C, RAD51D, RECQL, RECQL4, RECQL5, RPA1, WRN etc.

3. Small cell lung cancer that has progressed during or after first-line therapy.

* The 1st line regimen must have contained platinum-based regimen with or without iCPI.
* Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
* If the subject corresponds to sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), she / he should receive second-line treatment before entering the study 4. Subjects (male/female) must be > 18 years of age. 5. Subjects must have normal organ and bone marrow function measured within 14 days prior to administration of study treatment as defined below (transfusion allowed);
* Haemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* No features suggestive of MDS/AML on peripheral blood smear
* White blood cells (WBC) > 3x109/L
* Platelet count ≥ 100 x 109/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
* Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 51 mL/min (Cockcroft-gault method).

A. CrCl = (140-age) x (weight (kg)) x (0.85 for female) i. ---------------------------------------------------------- A. (72 x serum creatinine (mg/dL)) 6. ECOG performance status 0-2 subject must have a life expectancy ≥ 16 weeks. 7. Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Postmenopausal is defined as:

* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
* LH and FSH levels in the post-menopausal range for women under 50,
* radiation-induced oophorectomy with last menses > 1 year ago,
* chemotherapy-induced menopause with > 1-year interval since last menses,
* or surgical sterilization (bilateral oophorectomy or hysterectomy). 8. The subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

  9. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.

  10. Provision of informed consent for genetic research. 11. Male patients must use a condom during treatment and for 6 months after the last dose when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients and female patients should also use a highly effective form of contraception ([see appendix A for acceptable methods]) for 6 months after the last dose if they are of childbearing potential.

Exclusion Criteria:

1. Involvement in the planning and / or conduct of the study (applies to both AstraZeneca/Roche staff and / or staff at the study sites)
2. Previous enrolment in the any of SUKSES umbrella trials.
3. Participation in another clinical study with an investigational product during the last 2 weeks (or a longer period depending on the defined characteristics of the agents used).
4. Any previous treatment with a PARP inhibitor not limited to olaparib.
5. More than two prior chemotherapy regimens for the treatment of small-cell lung cancer. Pazopanib maintenance or immune checkpoint inhibitor (CTLA4, PD-1 or PD-L1 monoclonal antibody) is not considered as line of treatment.
6. Subjects with second primary cancer stable without treatment for 2 years are eligible for the trials. Adequately treated non-melanoma skin cancer, superficial urothelial tumor, early gastric cancer, in-situ cancer of the cervix, thyroid cancer or other solid tumours curatively treated with currently no evidence of disease is eligible for the trial.
7. Subjects receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The subject can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
8. Concomitant use of known CYP3A4 inhibitors.

   * Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting <<select olaparib or study treatment>> is 2 weeks
   * Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting <<select olaparib or study treatment>> is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
9. Persistent toxicities (> = CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
10. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Subjects with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The subject can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. The subjects with brain metastases who is previously treated and currently in stable status, no clinical symptom or image confirmed disease progression, are eligible for the trial. The subjects with untreated asymptomatic brain metastases is also allowed for the trial.
12. Major surgery within 14 days of starting study treatment or subjects not being recovered from any effects of any major surgery
13. Subjects considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled major seizure discorder, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression which cause neurologic symptom (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan which cause respiratory distress or any psychiatric disorder that prohibits obtaining informed consent.
14. Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Breastfeeding and pregnant women
16. Immunocompromised subject, e.g., subjects who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
17. Subjects with known active hepatic disease (i.e., Hepatitis B or C) due to the risk of transmitting the infection through blood or other body fluids.
18. Subjects with a known hypersensitivity to olaparib or any of the excipients of the product.
19. Subjects with uncontrolled seizures.
20. Exclusions related to bevacizumab

    * Inadequately controlled hypertension (defined as systolic blood pressure > 150mmHg and/or diastolic blood pressure > 100 mmHg) identified during the screening period and dose not resolved with resting or the treatment at the following measurement. (Patient can be re-screened after appropriate manage for lowering the blood pressure) Anti-hypertensive therapy to achieve these parameters is allowable.
    * Prior history of hypertensive crisis or hypertensive encephalopathy
    * Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
    * History of hemoptysis (one-half teaspoon of bright red blood per episode) within 1 month prior to randomization
    * Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
    * Current or recent (within 10 days of randomization) use of aspirin (325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
    * Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to randomization.

    The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the subject has been on a stable dose of anticoagulants for at least 2 weeks prior to randomization. The use of Direct Oral Anticoagulants is not recommended due to increased bleeding risk.

    Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR < 1.5 x ULN and aPTT is within normal limits within 14 days prior to randomization.

    Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
    * Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
    * History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to randomization
    * Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
    * Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
    * Serious, non-healing wound, active ulcer, or untreated bone fracture
    * Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection All subjects with ≥ 2 + protein on dipstick urinalysis at baseline must undergo a 24 hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours.
    * Known sensitivity to any component of bevacizumab
    * Clear tumor infiltration into the thoracic great vessels is seen on imaging
    * Clear cavitation of pulmonary lesions is seen on imaging
21. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation(dUCBT)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | through study completion, an average of 1 year
  Response rate of chemotherapy in patients.

SECONDARY OUTCOMES:
Overall survival (OS) and progression-free survival (PFS) | through study completion, an average of 1 year
  Patient survival and non-PD duration
Subgroup analyses based on biomarker | through study completion, an average of 1 year
  Analysis of treatment effects according to biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, Professor, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea